CLINICAL TRIAL: NCT04215549
Title: The Cost of Obsessive-compulsive Disorder (OCD) in China: Multi-center Cross-sectional Survey Based on Hospital
Brief Title: The Cost of Obsessive-compulsive Disorder (OCD) in China
Acronym: OCD
Status: Withdrawn | Type: Observational
Why Stopped: Because of COVID-19, we cann't carry out recruiting according to the original plan
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Capital Medical University (Other); Peking University Sixth Hospital (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Shandong Provincial Hospital (Other Government); Qingdao Mental Health Center (Unknown); the First Psychiatric Hospital of Harbin (Unknown); Qiqihar Medical University (Other); The Second Affiliated Hospital of Xinxiang Medical College (Unknown); Seventh People's Hospital of Hangzhou (Other); Guangji Hospital Affiliated to Soochow University (Unknown); First Affiliated Hospital of Kunming Medical University (Other); Brain Hospital Affiliated to Guangzhou Medical University (Unknown)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Other Study IDs: SMHC-OCD-5
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: OCD patients come from 13 hospitals located in the north, south, east and west of China
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — cross sectional study，no intervention

SUMMARY:
The purpose of this study is to estimate the cost of obsessive-compulsive disorder in China based on the prevalence rate from a social perspective.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder(OCD) is one of relatively common mental disorders with a prevalence of 1.63% in China. OCD usually begins in adolescence or young adulthood , it will become a chronic disabling disease, if it is not treated in timeand.OCD can be so severe that it can seriously impact on some or all areas of a person's life, bring huge economic burden. At present, there is only one article on the cost of OCD in the United States in the 1990s, and this part of the data in China is blank.A cross-sectional study recruited 600 patients with OCD from 13 hospitals in eastern, western, southern, and northern China. A structured questionnaire was used for face-to-face interviewing to collect costs related to OCD. The direct costs for each patient and indirect costs ffor each patient and their caregivers were calculated . The human capital method is used to calculate indirect costs. Through weighting, the cost of OCD in China is estimated from a social perspective using a bottom-up methodology.

ELIGIBILITY:
Inclusion Criteria:

* primarily diagnosed OCD meet DSM-5 critera
* 16-65 years old
* Get informed consent from patients

Exclusion Criteria:

* Concurrent neuropsychiatric diseases such as schizophrenia, which severely interfere with treatment costs
* Drug abuser
* Unable to understand the questionnaire

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with obsessive-compulsive disorder are recruited from both outpatient clinics and inpatient departments
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
obsessive-compulsive disorder related costs in China | 1 year
  Estimating the direct and indirect Costs of Chinese OCD based on prevalence from a social perspective

SECONDARY OUTCOMES:
Direct costs and indirect costs of consumed resources | 1 year
  Direct costs include medical costs and transportation, food, accommodation, etc. corresponding related to clinics.Indirect costs include lost time for patients and family members due to OCD.
other costs directly associated with OCD | 1 year
  Other medical costs and economic loss of disruptive behaviors due to OCD

CONTACTS AND LOCATIONS:
Overall Officials: Wang Zhen, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China